CLINICAL TRIAL: NCT06055725
Title: A Prospective, Multicountry Study to Estimate the Incidence of and Provide a Best Practice Model for Monitoring the Development of Post-Stroke Spasticity
Brief Title: A Study to Estimate How Often Post-stroke Spasticity Occurs and to Provide a Standard Guideline on the Best Way to Monitor Its Development
Acronym: EPITOME
Status: Recruiting | Type: Observational
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Other Study IDs: CLIN-52120-458
Record Dates: First submitted 2023-09-20; First posted 2023-09-28 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Spasticity as Sequela of Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study will monitor patients during the first year following their stroke.

Stroke is a very serious condition where there is a sudden interruption of blood flow in the brain.

The main aim of the study will be to find out how many of those who experience their first-ever stroke then go on to develop spasticity that would benefit from treatment with medication.

Spasticity is a common post-stroke condition that causes stiff or ridged muscles.

The results of this study will provide a standard guideline on the best way to monitor the development of post-stroke spasticity.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be aged 18 to 90 years at the time of providing informed consent
* First-ever clinical stroke, defined according to World Health Organization criteria as rapidly developing clinical signs of focal (at times global) disturbance of cerebral function lasting more than 24 hours, within the past 4 weeks;
* Confirmed paresis of the arms and/or legs which does not resolve within 1 day, according to the NIHSS score (a score of > 0 on Question 5 or 6 of the scale) within 2 weeks after the stroke
* Capable of giving informed consent which includes compliance with the requirements and restrictions listed in the ICF and in this protocol

Exclusion Criteria:

* Upper or lower extremity functional impairment prior to stroke per investigator judgement (e.g., modified Rankin Scale >2);
* Presence of significant/major neurological impairment that might affect muscle tone (other than limb paresis);
* Severe multi-impairment or diminished physical condition before stroke that could have caused paresis/spasticity/motor deficit per investigator judgement;
* Life expectancy of less than 12 months as a result of severity of stroke or other illnesses (e.g. cardiac disease, malignancy, etc.)
* Participation in any interventional study

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The Main Population will be participants aged 18 to 90 years with confirmed paresis within 2 weeks after a first-ever clinical stroke that has occurred within the past 4 weeks
Sampling Method: Non-Probability Sample
Enrollment: 1051 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2027-11-30 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants at the Clinical Confirmation Visit (CCV) who have problematic spasticity and who the investigator considers would benefit from pharmacological therapy | At the Clinical Confirmation Visit (CCV) up to maximum 18 months
  This is based on the investigator's clinical judgement and could include spasticity characterised by any of the following criteria aligned with the World Health Organization International Classification of Functioning, Disability and Health in three dimensions: Impairment, Activity limitations & Restriction on participation.

SECONDARY OUTCOMES:
Distribution of National Institutes of Health Stroke Scale (NIHSS) scores | At enrollment
  Including description of score for each physical item (arm and leg motor scores) and total physical item score National Institutes of Health Stroke Scale (NIHSS) is a 15-item impairment scale, intended to evaluate neurologic outcome and degree of recovery for patients with stroke. The scale assesses level of consciousness, extraocular movements, visual fields, facial muscle function, extremity strength, sensory function, coordination (ataxia), language (aphasia), speech (dysarthria), and hemi-inattention (neglect) (Lyden, Lu, & Jackson, 1999; Lyden, Lu, & Levine, 2001). The higher the NIHSS score the worse the outcome for the participant. If the participant has a score greater than '0' they will satisfy Inclusion Criteria number 3.
Percentage of participants who develop signs of possible spasticity | At Week 2, Month 1, Month 2, and every 3 months up to Month 12.
Percentage of participants who develop clinically confirmed spasticity | Week 2 to Month 14
Time from first ever stroke to detection of signs of possible spasticity | Week 2 to Month12
Time from first ever stroke to onset of clinically confirmed spasticity | Week 2 to Month 14
Time from first-ever stroke to onset of clinically confirmed problematic spasticity | Week 2 to Month 18
Description of signs of possible spasticity from the Post-stroke Spasticity Monitoring Questionnaire (PSMQ) | At Week 2, Month 1, Month 2, and every 3 months up to Month 12.
  Post-stroke Spasticity Monitoring Questionnaire (PSMQ) is a modified version (in local language) of a published 13-item patient reported screening questionnaire designed as a practical, easy-to-use tool to enable health care providers to identify patients with spasticity in need of treatment in routine clinical practice. The PSMQ will have an additional (14th) question for the participant to answer only if he/she has a total score for the first 13 questions of > 0 and has given an identical pattern of responses for any previously answered questionnaire which led to a F2F visit where a result of Modified Ashworth Scale (MAS) = 0 was obtained. The higher the PSMQ or MAS score is the worse the outcome for the participant.
MAS distribution at the CCV (overall and distribution by timing post-stroke) | Week 2 to Month 14
Distribution of spasticity (arm/leg, unilateral/bilateral, affected muscle groups) at the CCV | Week 2 to Month 14
Severity of spasticity by Modified Ashworth Scale (MAS) at the CCV | Week 2 to Month 14
MAS distribution (overall and distribution by timing post stroke) at the CCV | At Week 2, Month 1, Month 2, and every 3 months up to Month 14.
  MAS score per joint/muscle group and MAS total score by limb
MAS distribution of problematic spasticity at the CCV (overall and distribution by timing post-stroke) | Week 2 to Month 18
Distribution of problematic spasticity (arm/leg, unilateral/bilateral, affected muscle groups) Severity of problematic spasticity by MAS at the CCV | Week 2 to Month 18
Distribution of 36-Item Short-form Health Survey (SF-36) quality of life questionnaire scores in participants with clinically confirmed spasticity[c] at the CCV | Week 2 to Month 14
  Participants with clinically confirmed spasticity (MAS > 0 in any muscle group of arm and/or leg) at the CCV will be asked to complete the SF-36 health survey to assess their general health and wellbeing. The SF-36 is a generic, multipurpose short form survey consisting of 36 questions. Most of the questions are answered based on how the participant has been feeling over the previous 4 weeks.
Percentage of participants who develop problematic spasticity at the time of the confirmed diagnosis of spasticity at CCV | Week 2 to Month 14
Percentage of participants who develop problematic spasticity | At CCV and 4 months after the CCV
Stroke types | Week 2 to Month 14
  In terms of side (Left/Right), aetiology (Ischaemic/Haemorrhagic), and Bamford/Oxford classification (Total Anterior Circulation (TAC), Partial Anterior Circulation (PAC), Lacunar syndrome (LAC), Posterior Circulation syndrome (POC), occurrence of thrombolysis or thrombectomy.

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (58):
- United States (21):
  - Loma Linda, Anderson, California
  - University Of California, Los Angeles Medical Center, Los Angeles, California
  - University of South Florida (USF) - Morsani Center (USF Health Carol and Frank Morsani Center for Advanced Healthcare), Florida City, Florida
  - Knight Neurology, Rockledge, Florida
  - Emory University Merge, Atlanta, Georgia
  - Medstar Health Research Institute, Inc, Hyattsville, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Spaulding Rehabilitation Hospital, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - University of Missouri Health Care, Columbia, Missouri
  - Methodist Physicians Clinic, Omaha, Nebraska
  - Madonna Rehabilitation Hospital - Omaha Campus, Omaha, Nebraska
  - Duke University School of Medicine, Durham, North Carolina
  - Dayton Center for Neurological Disorders, Centerville, Ohio
  - Moss Rehab, Elkins Park, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - The University Of Texas Southwestern Medical Center, Dallas, Texas
  - McGovern Medical School - UT Physicians - Neurology (Adult Neurology Clinic) - Texas Medical Center Location, Houston, Texas
  - The University of Texas Health Science Center, San Antonio, Texas
  - University Of Utah, Salt Lake City, Utah
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- France (5):
  - CHU Bordeaux-Hopital Pellegrin, Bordeaux
  - CHU de Caen, Caen
  - CHU de Rennes, Hopital de Pontchaillou, Rennes
  - Hospices Civils de Lyon (HCL) - Hopital Henry Gabrielle, Saint-Genis-Laval
  - CHU Nantes, Saint-Jacques
- Germany (9):
  - Klinikum Altenburger Land GmbH, Altenburg
  - Charité - Universitaetsmedizin Berlin - Campus Charite Mitte (CCM), Berlin
  - University Hospital Carl Gustav Carus, Dresden
  - Heinrich-Heine-Universitaet Duesseldorf - Universitaetsklinikum Duesseldorf (UKD), Düsseldorf
  - Universitaetsklinikum Essen, Essen
  - Universitaetsklinikum Schleswig-Holstein, UKSH-Campus Kiel, Kiel
  - Universitaetsklinikum Schleswig-Holstein Campus Luebeck, Lübeck
  - Universitaetsmedizin der Johannes - Gutenberg Universitaet Mainz, Mainz
  - Universitaetsklinikum Tuebingen (UKT), Tübingen
- Italy (6):
  - Azienda Ospedaliero Universitaria OO RR di Foggia, Foggia
  - Milan University, Humanitas Clinical Institute, Milan
  - AOU maggiore della Carita', Novara
  - AOU San giovanni di Dio e Ruggi d'aragona Univ. di Salerno, Salerno
  - Neurological Rehabilitation Unit- Policlinico Borgo Roma., Verona
  - Neuromotor And Cognitive Rehabilitation Research Centre; Dep. Of Neurological, Neuropsychological, Morphological And Movement Sciences; Univ. Of Verona - Neurological Rehabilitation Unit- Policlinico Borgo Roma, Verona
- Spain (8):
  - Hospital Universitari Germans Trias i Pujol (HUGTP), Badalona
  - Hospital Mutua De Terrassa, Barcelona
  - Hospital Clinic i Provincial, Barcelona
  - Hospital Universitario La Paz, Madrid
  - Universidad Autonoma de Madrid (UAM) - Hospital Universitario de La Princesa, Madrid
  - Hospital Universitario Virgen del Rocio, Seville
  - Complexo Hospitalario Universitario De Vigo - Hospital Do Mexoeiro, Vigo
  - Hospital Universitario Miguel Servet de Zaragoza, Zaragoza
- Sweden (4):
  - Angelholm Northern Hospital, Ängelholm
  - Sodra Alvsborgs Sjukhus, Borås
  - Skane University Hospital, Malmo
  - Karnsjukhuset Skaraborg, Skövde
- United Kingdom (5):
  - University Hospitals of Leicester NHS Trust - Leicester General Hospital (LGH), Leicester
  - The Walton Centre, Liverpool
  - Kings College Hospital NHS Foundation Trust, London
  - South Tees Hospitals Foundation Nhs Trust, Middlesbrough
  - Nottingham University Hospitals NHS Trust - Nottingham City Hospital, Nottingham

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, annotated case report form, statistical analysis plan, and dataset specifications.
  Patient level data will be anonymized and study documents will be redacted to protect the privacy of study participants.
Time Frame: Where applicable, data from eligible studies are available 6 months after the studied medicine and indication have been approved in the US and/or EU.
Access Criteria: Further details on Ipsen's sharing criteria and process for sharing are available here (https://www.ipsen.com/science/clinical-trials/clinical-data-transparency/).
URL: https://www.ipsen.com/science/clinical-trials/clinical-data-transparency/

REFERENCES:
- [Derived] Zorowitz RD, Barrenechea LS, Butet S, Groppa S, Hernandez Herrero D, Prasad R, Sandars S, Meloni S, Page S, Maisonobe P, Picelli A. How many stroke survivors develop problematic spasticity requiring pharmacological therapy? An international (Europe and USA) observational study protocol. BMJ Open. 2025 Jan 15;15(1):e087404. doi: 10.1136/bmjopen-2024-087404. PMID 39819949